CLINICAL TRIAL: NCT04976426
Title: Establishment and Clinical Validation of a New Technique for Early Diagnosis of Diabetic Nephropathy
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Second Affiliated Hospital of Wenzhou Medical University (Other); Lishui Country People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: zhengchao3
Record Dates: First submitted 2021-06-24; First posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus; Biomarkers; Diabetic Kidney Disease; Early Diagnosis
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Nephropathies; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diabetic kidney disease(DKD) is a leading cause of chronic kidney disease and end-stage renal disease across the world. Early identification of DKD is vitally important for the effective prevention and control of it. However, the available indicators are doubtful in the early diagnosis of DKD. This study aims to develop a novel system of multidimensional network biomarkers (MDNBs) to estimating early diabetic nephropathy, and further validating the performance of the novel systemin in prediction of the risk for early diabetic nephropathy by a nested case-control study.

DETAILED DESCRIPTION:
Patients with a history of more than 5 years of diabetes without DKD were recruited. At the baseline visit, the patients' serum, plasma and urine were collected after obtaining informed patient consent. Simultaneously, the basic information, anthropometric indicators (including height, weight, waist circumference, hip circumference, blood pressure), past history, family history, menstrual history, birth history, medication history, lifestyle of the patients were registered, and the corresponding laboratory examination and auxiliary examination were carried out according to the diagnostic process. All data and data were entered into the database for later analysis. After 5years of follow up, subjects will be divided into two groups(the new onset DKD group and the non-DKD group), the base line level of MDNBs were tested in the two group to validate the performance of the novel MDNBs in in prediction of the risk for early diabetic nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have signed informed consent.
* Subjects who were diagnosed with diabetes at least 5 years.
* Subjects showed good compliance, and the follow-up data was available for >5 years.

Exclusion Criteria:

* Renal diseases caused by other causes, including primary and secondary;
* All kinds of acute infections;
* The expected life expectancy (life expectancy or related diseases) was less than 5 years according to the researcher's judgment.
* Drug users or drug abusers;
* Sexually transmitted diseases such as viral hepatitis, AIDS and syphilis, and infectious diseases such as tuberculosis are in an active period;
* Any situation judged by the researcher that affects enrollment.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The diagnosis of T2DM in our study complied with the criteria set out by the American Diabetes Association. The inclusion criteria are as follows: for all patients diagnosed with T2DM without CKD. After five years of following up，participants were recruited and then divided into two groups: T2DM group without nephropathy(non-DKD, UACR urinary albumin/creatinine ratio < 3 mg/mmol) and DKD group with microalbuminuria and macroalbuminuria (DKD, UACR > 3 mg/mmol)
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
multidimensional network biomarkers | 5years
  a novel system of multidimensional network biomarkers (MDNBs) based on a widely targeted metabolomics. Our previous study demonstrated that the combination of Linolelaidic Acid (C18:2N6T), L-Dihydroorotic Acid, and Azoxystrobin Acid might serve as a potential multidimensional network biomarkers of DKD. So we create a panel of MDNBs containing these biomakers as primary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Chao, MD, PhD, Principal Investigator — the Second Affiliated Hospital Zhejiang University Schoolof Medicine

IPD SHARING:
Plan to Share IPD: No